CLINICAL TRIAL: NCT05410015
Title: Evaluation of Prognostic Monitoring for Women Who Have Completed Standard Via Analysis of Immunoinflammation-related Protein Complexes in Blood
Brief Title: Evaluation of Prognostic Monitoring for Women Who Have Completed Standard Treatment for Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-OC1
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 mL of serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Normal clinical treatment without intervention — Normal clinical treatment without intervention

SUMMARY:
The relationship between immune inflammation-related protein complexes inblood and recurrence or metastasis of ovarian cancer will be studied

DETAILED DESCRIPTION:
100 cases in normal ovarian control group, 100 cases in benign ovarian disease group and 100 cases in malignant ovarian epithelial carcinoma group will be studied. Change regularity of ovarian cancer specific immune inflammation-related protein complexes in blood will be studied. The relationship between disease-specific protein complexes and pathological state of patients will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Normal ovary control
* Ovarian benign disease
* Ovarian malignant epithelial carcinoma

Exclusion Criteria:

* Male
* Age above 70
* Suffering from other malignant tumors
* Non-compliant patient

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population included normal ovarian controls, patients with benign ovarian disease, and patients with malignant epithelial ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Immune Inflammation-Related Protein Pomplexes | 2 years
  The change of immune inflammation-related protein complexes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No